# **Informed Consent**

**Date: 15-August-2024** 

**Title:** Efficacy of Psychological Intervention in Children with Cancer: A Randomized Controlled Trial (RCT)

**Principal Investigator (PI):** Dr. Muhammad Waseem Khan (Post Graduate Trainee)

Institution: Pediatric Oncology Unit, The Children's Hospital, PIMS Islamabad, Pakistan

#### **Introduction:**

We invite you to participate in a research study aimed at evaluating the effectiveness of a psychological intervention in improving the mental health and well-being of children with cancer. Your participation will help us better understand how to support children with cancer and their families.

## **Purpose:**

The purpose of this study is to evaluate the efficacy of a psychological intervention in reducing symptoms of anxiety, depression, and post-traumatic stress disorder (PTSD) in children with cancer.

#### Procedure:

If you agree to participate, your child will be randomly assigned to either the intervention group or the control group. The intervention group will receive a psychological intervention consisting of cognitive-behavioral therapy and relaxation techniques. The control group will receive standard care. Your child's participation will involve \_\_\_\_\_\_ sessions of \_\_\_\_\_ each.

#### **Risks and Benefits:**

There are no anticipated risks associated with this study. The potential benefits include improved mental health and well-being for your child.

## **Confidentiality:**

Your child's personal and medical information will be kept confidential and stored securely.

### **Voluntary Participation:**

Your participation is voluntary, and you may withdraw your child from the study at any time without penalty.

### **Contact Information:**

If you have any questions or concerns, please contact Dr. Muhammad Wasim Khan at 0333-4411620 or 051-90714250.

| Consent: | |
|---|---|
| | , hereby provide informed consent for my child,<br>idy. I understand the purpose, procedure, risks, and benefits, a<br>participate. |
| Signature: | |
| Date: | _ |
| Time: | |